CLINICAL TRIAL: NCT05300711
Title: Preventing Ovarian Cancer Through the Expansion of Opportunistic Salpingectomy: Uptake, Safety and Cost-effectiveness at the Time of Colorectal Surgery
Brief Title: Preventing Ovarian Cancer Through Oportunistic Salpingectomy at the Time of Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Gillian Hanley, Assistant Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H22-003399
Record Dates: First submitted 2022-02-23; First posted 2022-03-29 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Salpingectomy; Colorectal Surgery
Keywords: Salpingectomy; Colorectal Surgery; Ovarian Neoplasms; Primary Prevention
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opportunistic salpingectomy (Experimental): The participating surgeons will attempt to perform bilateral salpingectomy in addition to the colorectal surgery.
  Interventions: Procedure: Bilateral salpingectomy; Procedure: Colorectal surgery
- Colorectal surgery only (Active Comparator): Participants will receive the standard of care, that is colorectal surgery.
  Interventions: Procedure: Colorectal surgery

INTERVENTIONS:
Procedure: Bilateral salpingectomy — Removal of both fallopian tubes.
  Arms: Opportunistic salpingectomy
Procedure: Colorectal surgery — Colorectal surgery as indicated by attending surgeon.

SUMMARY:
This study aims to evaluate the feasibility, safety and cost-effectiveness of opportunistic salpingectomy (OS-the removal of the fallopian tubes) at the time of colorectal surgery to prevent ovarian cancer. Ovarian cancer is the fifth cause of cancer-related mortality in females in Canada. OS can prevent the most common and lethal type of ovarian cancer, high grade serous carcinoma (HGSC). OS during gynecologic surgery (hysterectomy or instead of tubal ligation) is safe and effective. However, rates of hysterectomies and tubal sterilization are decreasing. This research team aims to extend the prevention of ovarian cancer by expanding to offer OS during other surgeries in the pelvis where fallopian tubes are accessible, beginning with colorectal surgery. This study will examine: 1) the feasibility of OS at the time of colorectal surgery; 2) the safety of OS at the time of colorectal surgery; 3) the cost-effectiveness of OS at the time of colorectal surgery.

The hypothesis is that OS will be well accepted by individuals with fallopian tubes undergoing colorectal surgery, and that the vast majority (around 90 percent) of attempts to remove both fallopian tubes will be successful. It is expected that there will be 10-20 minutes additional operating room time for completing OS and that there will be no increased risk of complications when OS is included in a colorectal surgery. The researchers also hypothesize that OS at the time of colorectal surgery will be cost-effective because of the reduced number of ovarian cancer cases and associated treatment costs.

DETAILED DESCRIPTION:
Research design:

120 eligible participants will be enrolled and consented to undergo OS at the time of colorectal surgery. As a control group, 120 participants undergoing colorectal surgery without OS will be included. When eligible participants decline OS, they will be approached to participate as a control, and once 120 participants have consented to OS, participants will be enrolled as controls until there are 120 patients in the control group.

Methods and analysis:

The research coordinator will contact participants to consent them to undergo OS or to participate as a control participant at a preoperative visit prior to their colorectal surgery. The research coordinator will walk them through the informed consent form and answer any questions about the study. This will occur either at St Paul's Hospital, or over the phone or via telehealth video conference.

Information will be collected regarding all participants who were approached to consent for OS. For those who agree to participate in the study, a short questionnaire will be applied to collect some additional information that would not be available in the chart. Those who decline OS will be asked about their reasons for not participating to better understand the patient perspective, inform future research and develop lay communication materials around OS. The percentage of participants who consented to OS will be calculated, as well as those who successfully had both fallopian tubes removed during their colorectal surgery.

To calculate how much additional operating room (OR) time is required when OS is performed concurrently with colorectal surgery, the research coordinator will attend the OR and record the amount of time taken for both fallopian tubes to be removed or for the attempt to be abandoned (in rare cases where both tubes are not removed).

To assess the safety of providing OS at the time of colorectal surgery, postoperative complications will be addressed, including duration of hospital stay and 30-day hospital readmission rate, blood transfusion and surgical site infection. All participants will receive standard post-operative care. All data on perioperative complications are available in the participant's medical chart. The research coordinator will access this information for the research team. Perioperative complications will be graded according to the Clavien-Dindo classification of surgical complications, which uses a grading approach. Grade 1 represents any deviation from the normal postoperative course that does not require the need for additional treatment beyond the use of antiemetics, antipyretics, analgesics, diuretics, electrolytes and physiotherapy. Grade 2 represents complications that require pharmacologic treatment beyond what is included for grade 1 complications and includes blood transfusions. Grade 3 includes complications that require surgical, endoscopic, or radiological intervention, Grade 4 includes life threatening complications requiring admission to intensive care and Grade 5 is death of the patient.

To determine the cost effectiveness of OS at the time of colorectal surgery, the data generated regarding additional OR time and any additional complications will be used to conduct Markov Monte Carlo simulation models. Monte Carlo simulations will estimate the number of people who will be diagnosed with HGSC in the future after OS compared to those not having this procedure, based on the effectiveness data generated from OS at the time of hysterectomy and tubal ligation. Direct and indirect health care costs will be derived from previously existing sources, including patient cost estimators from the Canadian Institute for Health Information that includes provincial cost estimates for colorectal surgeries by province. Lifetime risks of HGSC will be modeled from the Canadian Cancer Statistics. Competing mortality risks that are age and sex dependent will be derived from Canadian Life Tables. The researchers will use published costs for treatment of HGSC and compare the direct HGSC-related costs (costs associated with either prevention or treatment of HGSC) across the groups.

Reporting for adverse events:

All potential side effects related to study interventions will be recorded. Adverse events will be monitored on an ongoing basis by the research coordinator, and frequencies will be reported to investigators bimonthly.

Any Clavien-Dindo complication of 3, 4, or 5 (more serious) will be immediately reviewed. The rate of Clavien-Dindo grade 1 and 2 complications will be reviewed at interim analyses, which will be conducted when 1/3 of participants have been recruited and again when 2/3rd have been recruited.

If the study shows that adverse events, serious or not, are occurring at a higher rate for people undergoing OS compared to baseline expected rates the study may be stopped early. If unanticipated adverse events are discovered, the study may be stopped early. In either case, there would be no further recruitment.

In the case of study stoppage, all colorectal surgeons at St Paul hospital will be immediately notified in writing. The research coordinator will no longer recruit and consent patients at St Paul's hospital.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with intact fallopian tubes.
* Individuals undergoing one of the following open or laparoscopic colorectal surgery: total colectomy, right hemicolectomy, left hemicolectomy, anterior resection, low anterior resection, small bowel resection and appendectomy.
* Individuals who finished with childbearing.

Exclusion Criteria:

* Presence of BRCA 1 or 2 mutation.

Ages: 15 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The percentage of participants who consented to OS | When the patient is approached and asked to consent and when they decline or consent (~2-4 weeks)
  The percentage of participants who were approached who ultimately consented
The percentage of the participants who consented to OS who had both fallopian tubes removed. | During the surgical intervention (~2 hours for surgical intervention)
  The percentage of participants who consented and underwent removal of both fallopian tubes at the time of their surgery.
The number of additional minutes in the OR required to attempt or complete opportunistic salpingectomy during colorectal surgery (on average) | During the surgical intervention, a stopwatch will be started when fallopian removal begins and stopped when it is complete (~20 minutes)
  Average number of minutes spent removing fallopian tubes or attempting to remove fallopian tubes in the situation where removal of both tubes is unsuccessful.
Incidence of treatment emergent adverse events as assessed by the Clavien Dindo Clavien-Dindo classification of surgical complications. | These will be assessed during the surgical intervention and the 30 days following the surgical intervention.
  Rate of surgical complications among participants undergoing OS at the time of colorectal surgery compared with a control group of patients undergoing colorectal surgery without OS.

SECONDARY OUTCOMES:
Cost-effectiveness of OS as measured by the cost per quality adjusted life year | Following study completion; an average of 2 years
  We will calculate the cost per quality adjusted life year of performing OS at the time of colorectal surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Hanley, PhD, Principal Investigator — University of British Columbia; Heather Stuart, MD, Principal Investigator — University of British Columbia; Carl Brown, MD, Principal Investigator — St. Paul's Hospital
Locations (2):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No